CLINICAL TRIAL: NCT01483586
Title: Efficacy and Safety of Oral Kanglaite (KLTc)in Men With Prostate Cancer: Randomized, Dose-Ranging Study of the Effects of KLTc on Prostate Specific Antigen (PSA) Doubling Time Among Men With Rising PSA Levels After Definitive Local Therapy
Brief Title: Safety and Efficacy of Kanglaite Gelcaps in Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: KangLaiTe USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C10-069
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KLTc high dose (Experimental): 6 KLTc gelcaps taken four times a day
  Interventions: Drug: Kanglaite gelcap
- KLTc low dose (Experimental): 3 KLTc gelcaps taken four times a day
  Interventions: Drug: kanglaite gelcap

INTERVENTIONS:
Drug: kanglaite gelcap — 3 KLTc gelcap capsules four times a day throughout the study (12 months). Each gelcap contains .45g KLT per capsule
  Arms: KLTc low dose
Drug: Kanglaite gelcap — 6 KLTc gelcaps taken four times a day throughout the study (12 months). Each gelcap contains .45g KLT
  Arms: KLTc high dose

SUMMARY:
This research is being done to evaluate the safety and efficacy of the investigational Kanglaite gelcap (KLTc) on PSA in men with prostate cancer when given for twelve months.

ELIGIBILITY:
Inclusion Criteria:

* confirmed adenocarcinoma of the prostate
* undergone definitive treatment (surgery, surgery with radiation therapy, cryotherapy, radiation therapy or brachytherapy) for the primary prostate tumor with a rising PSA
* life expectancy greater than 6 months
* has Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* use of other dietary/herbal supplements (e.g. saw palmetto, selenium, etc.) has been stable for at least 2 months prior to screening and the patient agrees not to stop or change the dose while participating in the study.
* Adequate hepatic function with serum bilirubin ≤ 1.5 times the upper institutional limits of normal, ALT and AST ≤ 2.5 times the upper institutional limits of normal
* Adequate renal function with serum creatinine ≤ 1.5 times the upper institutional limits of normal
* Adequate hematologic function (absolute neutrophil counts ≥ 1,500 mm3 and platelets ≥ 100,000 mm3)
* All electrolytes (including potassium, sodium, and serum or ionized calcium) must be within normal limits

Exclusion Criteria:

* Patients with evidence of metastatic disease would be excluded, except for presence of positive lymph nodes from the surgical pathology. Similarly, patients with radiological evidence of lymph nodes < 2 cm that lack pathological confirmation would be eligible
* Patients with a PSA doubling time of <6months at screening would be excluded
* Patients meeting Phoenix criteria for biochemical failure (nadir + ≥2ng/mL increase in serum PSA) who wish additional conventional therapy
* Any concurrent malignancy other than adequately treated basal or squamous cell skin cancer or superficial bladder cancer
* Any psychiatric or other disorders such as dementia that would prohibit the patient from understanding or rendering informed consent or from fully complying with protocol treatment and follow-up
* Inability to swallow capsules
* Patients with a known history of gastrointestinal disease, surgery or malabsorption that could potentially impact the absorption of the study drug
* Patients requiring the use of a feeding tube
* Receipt of prior chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
prostate specific antigen doubling time (PSADT) | over 12 months on study drug
  PSADT is defined as the natural log of 2 (0.693)divided by the slope (beta- rate of change) of the relationship between the log of PSA and the time of PSA measurement using linear regression model

SECONDARY OUTCOMES:
PSA objective response | over 12 months on study drug
  a 50% or more decline in PSA level compared to baseline
KLTc intake compliance | each month, up to 12 months on study drug
  actual number of capsules taken divided by the expected number of capsules taken multiplied by 100 to get a percentage of compliance

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - North Shore University, Evanston, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina